CLINICAL TRIAL: NCT04360707
Title: Clinical Presentation and Incidence of SARS-CoV-2 Infection in Different Cohorts of Solid Organ Transplant Patients and Follow-up in France
Brief Title: Solid Organ Transplant Recipients With SARS-CoV-2 French Registry
Acronym: TX-COVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7766
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: SARS-CoV-2
Keywords: SARS-CoV-2; Covid-19; Solid Organ transplantation; Incidence; Prognosis; Cellular response; Humoral Response
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with comorbid condition are known to be at high risk of severe forms of Covid-19. It is highly probable that immunocompromised patients like solid organ transplant (SOT) recipients are also at risk of severe forms of Covid-19. For this purpose, The investigators conducted a nationwide multicentric and multiorgan Registry to collect data about all French SOT recipients who develop a SARS-CoV-2 infection. The aim is to describe the clinical, biological and virological characteristics of these patients and to give information about evolution and prognosis of these particular population

ELIGIBILITY:
Inclusion Criteria:

* All Solid Organ Transplant recipients with a functioning graft and a high suspicion or a confirmed SARS-CoV-2 infection
* Adult and pediatric

Exclusion Criteria:

- There are no exclusion criteria, except for the patient's explicit refusal to participate

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Solid Organ Transplant recipients with a functioning graft and a high suspicion or a confirmed SARS-CoV-2 infection
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-04-08 (Actual); Primary Completion 2021-04-08 (Estimated); Study Completion 2021-04-08 (Estimated)

PRIMARY OUTCOMES:
Clinical Presentation and Incidence of Covid-19 Infection in Different Cohorts of Solid Organ Transplant Patients | From 1st March 2020 to 1st March 2021

CONTACTS AND LOCATIONS:
Overall Officials: Sophie CAILLARD, MD, PhD, Study Director — Service de Néphrologie et Transplantation
Locations (1):
- Service de Néphrologie et Transplantation, Strasbourg, France

REFERENCES:
- [Derived] Gerard AO, Barbosa S, Anglicheau D, Couzi L, Hazzan M, Thaunat O, Blancho G, Caillard S, Sicard A; French SOT COVID Registry. Association Between Maintenance Immunosuppressive Regimens and COVID-19 Mortality in Kidney Transplant Recipients. Transplantation. 2022 Oct 1;106(10):2063-2067. doi: 10.1097/TP.0000000000004254. Epub 2022 Jul 27. PMID 35883236